CLINICAL TRIAL: NCT06125366
Title: Randomized, Single-blind, Placebo-controlled, Escalating Single-dose Study to Investigate Safety, Tolerability, and Pharmacokinetics of Intravenously Administered BAY 1747846 in Japanese Healthy Male Subjects
Brief Title: A Study to Learn More About the Safety and the Level of BAY 1747846 in Body Given as Injection Into the Vein at Increasing Single Doses in Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 19414
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging; Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study is performed according to a single-blind design, i.e. the participant is blinded to the allocation of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation of BAY1747846 (Experimental)
  Interventions: Drug: BAY1747846
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: BAY1747846 — Single dose; IV injection.
  Arms: Dose escalation of BAY1747846
Drug: Matching placebo — Single dose; IV injection.
  Arms: Matching Placebo

SUMMARY:
The goal of this clinical study was to learn more about BAY1747846 compared to placebo when given as an injection into the vein in Japanese healthy male participants:

* the safety of BAY1747846 when given at increasing single doses
* the level of BAY1747846 in the body over time when given at increasing single doses.

To answer the first question, the researchers compared the number and severity of medical problems the Japanese participants had after receiving BAY 1747846 at increasing doses and placebo respectively. Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

To answer the second question, the researchers determined:

* the (average) total level of BAY1747846 in the body, also called AUC
* the (average) highest level of BAY1747846 in the body, also called Cmax
* how BAY1747846 is removed from the body, also called clearance (CL).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study specific tests or procedures
* Ability and willingness to understand and follow study-related instructions
* Subject is healthy as determined by the investigator
* Japanese male
* Age 20 to 40 years (inclusive) at screening visit
* Body mass index (BMI): 18.0 to 28.0 kg/m^2(inclusive)
* Body weight: at least 50 kg (inclusive)
* Subjects of reproductive potential must agree to use condoms whenever having sexual intercourse with a woman of child-bearing potential. This applies to the time period from signing of the ICF to at least 1 week after treatment.

Exclusion Criteria:

* Current smoker, or has smoked within 3 months prior to screening Clinical Study Protocol
* Any severe disease within the last 4 weeks prior to administration of study drug
* History of orthostatic hypotension, fainting spells and blackouts
* Any malignant tumor and history thereof
* Any clinically relevant finding at the physical examination
* Any known disposition for allergic, anaphylactoid, hypersensitivity or idiosyncratic reactions, e.g. any history of clinical signs of hypersensitivity reaction to any contrast agent
* Any clinically relevant deviation from reference ranges of the laboratory parameters at screening or alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin exceeding the Upper limit of normal range (ULN) by more than 10%, or creatinine above the ULN, or hemoglobin below 12 g/dL
* Clinically relevant ECG findings, e.g.: Heart rate <45 or > 90 beats/min, PR >220 msec, QTcF >450 msec, QRS >120 msec, branch bundle block, any sign of coronary heart disease at screening

  -. Abnormal vital signs, e.g.: Systolic blood pressure <90 or >140 mmHg, Diastolic blood pressure <45 or >90 mmHg at screening
* Subjects who have participated in a clinical study of an investigational drug within 4 months or an approved drug within 3 months prior to administration of study drug

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events | Up to 7 to 10 days after study drug administration (From the time of signing of the ICF until the last visit of follow-up.)
Severity of treatment-emergent adverse events | Up to 7 to 10 days after study drug administration (From the time of signing of the ICF until the last visit of follow-up.)

SECONDARY OUTCOMES:
Maximum observed drug concentration in measured matrix after single dose administration (Cmax) | Pre-dose, on Day 1, Day 2, Day 3 and Day 4.
Area under the concentration vs. time curve from zero to infinity after single dose (AUC) | Pre-dose, on Day 1, Day 2, Day 3 and Day 4.
Total body clearance of drug (CL) | Pre-dose, on Day 1, Day 2, Day 3 and Day 4.
Total body clearance of drug normalized by body weight (CL/bw) | Pre-dose, on Day 1, Day 2, Day 3 and Day 4.

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/19414